CLINICAL TRIAL: NCT02991820
Title: Comparison of Miller and Macintosh Laryngoscopes, CMAC and Glidescope Videolaryngoscopes in Inexperienced Users: a Pediatric Manikin Study
Brief Title: VL vs DL in Inexperienced Users: a Pediatric Manikin Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: IRB16-00549
Record Dates: First submitted 2016-12-06; First posted 2016-12-14 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Videolaryngoscopes (VL); Direct Laryngoscopy (DL); Inexperienced Users

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inexperienced users (Experimental): Inexperienced users will include trainees (SRNAs, residents, fellows, and medical students) and nurses at NCH.
  Interventions: Device: Miller; Device: Macintosh; Device: C-MAC; Device: GlideScope
- Experienced users (Experimental): Experienced users will include faculty pediatric anesthesiologists CRNAs.
  Interventions: Device: Miller; Device: Macintosh; Device: C-MAC; Device: GlideScope

INTERVENTIONS:
Device: Miller — Direct laryngoscopy and endotracheal intubation attempted by each provider using direct laryngoscopy (DL) with a Miller laryngoscope
Device: Macintosh — Direct laryngoscopy and endotracheal intubation attempted by each provider using DL with a Macintosh laryngoscope
Device: C-MAC — Indirect laryngoscopy and endotracheal intubation attempted by each provider using the C-MAC video laryngoscope
Device: GlideScope — Indirect laryngoscopy and endotracheal intubation attempted by each provider using the GlideScope video laryngoscope

SUMMARY:
This study will compare the CMAC and Glidescope videolaryngoscopes (VL) to traditional direct laryngoscopy (DL) using either a Miller or Macintosh laryngoscope by studying the performance of users. This will involve the use of an intubating pediatric manikin to assess various aspects of endotracheal intubation by experienced and inexperienced users.

DETAILED DESCRIPTION:
The commonly used method for endotracheal intubation in children is direct laryngoscopy using a Miller or Macintosh blade. Videolaryngoscopy is a widely accepted pediatric airway management. Videolaryngoscopes (VL) provide an indirect view of glottis without the need to align the oral, pharyngeal, and glottis structures. Some types of VLs provide also direct view of glottis with indirect view. Videolaryngoscopes can be used as a teaching tool for learners as they can visualize all the anatomical structures of larynx at the same time with the performer. VLs may facilitate the learning of endotracheal intubation in inexperienced users in the pediatric population. There are limited data on the use of videolaryngoscopes by anesthesia providers and medical personnel who are inexperienced in the use of videolaryngoscopes.

ELIGIBILITY:
Inclusion Criteria:

* Faculty pediatric anesthesiologists
* CRNAs
* Trainees (SRNAs, residents, fellows, and medical students)
* Nurses from NCH

Exclusion Criteria:

* If subjects are unwilling to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Inexperienced Users: Inexperienced users will include trainees (SRNAs, residents, fellows, and medical students) and nurses at NCH.
  Intubation: Each participant will perform endotracheal intubation on the mannequin using videolaryngoscopes (VL) and traditional direct laryngoscopy (DL).
- Experienced Users: Experienced users will include faculty pediatric anesthesiologists CRNAs.
  Intubation: Each participant will perform endotracheal intubation on the mannequin using videolaryngoscopes (VL) and traditional direct laryngoscopy (DL).
Period: Overall Study
Arm/Group | Inexperienced Users | Experienced Users
Started | 12 | 31
Completed | 12 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inexperienced Users | Experienced Users | Total
Number analyzed (Participants) | 12 | 31 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 31 | 43
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — was not assessed | NA — was not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — was not assessed | NA — was not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 31 | 43

OUTCOME MEASURES:

1. Primary Outcome: Time to Endotracheal Intubation
Description: The amount of time it took to successfully intubate the manikin using each device.
Time Frame: the same day (within seconds to minutes)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Inexperienced Users | Experienced Users
Number analyzed (Participants) | 12 | 31
seconds
  Miller | 72 (45) | 30 (28)
  Macintosh | 72 (45) | 27 (23)
  C-Mac | 61 (34) | 20 (13)
  GlideScope | 118 (6) | 85 (38)

2. Secondary Outcome: Successful Intubation Within 120 Seconds
Description: The number of participants who were able to successfully intubate the manikin using each device within 120 seconds.
Time Frame: 2 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Inexperienced Users | Experienced Users
Number analyzed (Participants) | 12 | 31
Participants
  Miller | 7 | 30
  Macintosh | 7 | 31
  C-Mac | 11 | 31
  GlideScope | 2 | 20

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Inexperienced Users | Experienced Users
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT02991820/Prot_SAP_000.pdf